CLINICAL TRIAL: NCT06705920
Title: Effect of Topical Active Oxygen Therapy on Surgical Site Wound Healing and Microbial Colonization : Randomized Controlled Clinical Trial
Brief Title: Effect of Topical Active Oxygen Therapy on Surgical Site Wound Healing and Microbial Colonization
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: British University In Egypt (Other)
Responsible Party: Principal Investigator, ahmed hamdy mahmoud, assistant lecturer, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-042
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Patients Scheduled for Any Oral Surgical Flap Procedure That Require Suturing Will Be Included in This Study
Keywords: active oxygen; sutures; flap; microbiology; wound healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): patient who will undergo intraoral surgical procedures , will have his wound sutured without any addtives
- test (Active Comparator): patient who will undergo intraoral surgical procedures , will have his wound sutured with the addition of blue m gel twice daily
  Interventions: Drug: topical oxygen gel

INTERVENTIONS:
Drug: topical oxygen gel — In the study group the gel will be applied over the suture and the patients will be instructed to apply the gel to the wound area and to the suture thread using a cotton swab
  Arms: test

SUMMARY:
To assess the antibacterial efficiency of oxygenated gel therapy on wound healing and microbiological colonization around surgical sutures

DETAILED DESCRIPTION:
All the patients who will agree to participate in the study and who will sign the informed consent forms. Computer-generated randomization will be used to randomly divide the surgical sites into two groups. Control group: will receive no treatment. Study group: will receive active oxygen gel around suture. Patients scheduled for any oral surgical flap procedure that require suturing will be included in this study. After flap approximation, the surgical site will be sutured using 5-0 braided sutures. In the study group the gel will be applied over the suture and the patients will be instructed to apply the gel to the wound area and to the suture thread using a cotton swab, three times a day after brushing their teeth. Also, patients will be given instructions regarding their post-surgical care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients in a healthy systemic condition who required comprehensive dental treatment
* Both genders with age group > 18 years old
* Patients should approve to deliver a signature to a written consent after study nature explanation.

Exclusion Criteria:

* Patients with severe smoking habits >10 cig \ day
* Pregnant females, decisional impaired individuals and handicapped patients
* Patients having poor oral hygiene or not wanting to carry out oral hygiene measures
* Patients on any medication affecting the soft tissue health (e.g., amlodipine, Cyclosporine A, hydantoin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Post operative wound healing. | 2 weeks
  Wound healing will be recorded in the 1st and 2 weeks postoperatively through Landry Wound Healing Index (LWHI) which evaluates the surgical site based on tissue color, response to touch, the marginality of the incision line, and extent of the area. The rating is from 1 = very poor to 5 = excellent.

SECONDARY OUTCOMES:
Microbiological assessment | 2 weeks
  The collected samples of suture thread will be immersed in phosphate-buffered saline solution (PBS) immediately after their removal and This sample will be subsequently sent to the microbiology laboratory of the Faculty of Pharmacy of the British university in Egypt. The samples will be shaken vigorously for two minutes to separate the bacteria from the suture thread, and to obtain a homogeneous suspension. serial dilutions in saline will be subsequently prepared. 50 microliters of each dilution will be plated in Petri dishes containing different culture media.The blood agar, mannitol agar, MacConkey agar, and Sabouraud agar plates will be aerobically incubated at 37 °C for 24-48 hours. After incubation, the colony forming units (CFUs) will be counted and the total number of CFUs per milliliter of initial solution will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Sherouk, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol